CLINICAL TRIAL: NCT06216457
Title: Study on the Performance of a Machine Learning Algorithm Recognizing and Triaging Large Vessel Occlusions Using Non-contrast CT Scans
Acronym: SMART-LVO
Status: Not yet recruiting | Type: Observational
Sponsor: Methinks Software SL (Industry)
Collaborators: Santiago Ortega- global PI (Unknown)
Responsible Party: Sponsor
Other Study IDs: SMART-LVO Registry
Record Dates: First submitted 2024-01-04; First posted 2024-01-22 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic; Stroke, Acute; Brain Ischemia
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Stroke; Brain Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Group 1: LVO: Subjects with Methinks NCCT algorithm detecting ICA, M1, and M2 occlusions.
  Interventions: Device: AI software for Stroke
- Group 2: ICH: Subjects with Methinks NCCT algorithm detecting ICHs.
  Interventions: Device: AI software for Stroke
- Group 3: Controls: Subjects with final diagnosis confirmed not to be Stroke (i.e. stroke mimic) or any type of stroke not determined to be: LVO (ICA, M1 or M2) or ICH.
  Interventions: Device: AI software for Stroke

INTERVENTIONS:
Device: AI software for Stroke — AI Software for Non-Contrast Head CT (Computed Tomography) and CT Angiography, utilized for Code Stroke screening, notification and triage.
  Other Names: Methinks AI Software

SUMMARY:
The goal of this prospective observational study is to assess the effectiveness and performance of Methinks AI stroke imaging software platform in acute Code Stroke patients, and as a comparator to study sites utilizing existing AI imaging stroke platforms.

The main question[s] it aims to answer is:

• Performance of and outcomes associated with the use of the Methinks AI stroke imaging medical device in real-world clinical practice.

DETAILED DESCRIPTION:
This is a prospective observational medical device clinical trial that aims to assess the diagnostic performance of Methinks Investigational Device on detecting LVO and ICH on plain NCCT and CTA, in consecutive acute Code Stroke activations at the emergency department.

Demographic, Clinical and Imaging variables will be collected from stroke onset through Day 7 or Discharge, whichever is earlier. Methinks results will be collected exclusively for research purposes and no clinical decisions will be made based on the output. Diagnostic performance of NCCT-LVO Methinks output will be assessed using DSA and/or CTA as ground truth. Presence of ICH will be assessed using an independent neuroradiologist final reading. The Clinical impact on workflow will be retrospectively estimated based on the reduction of time to decision in both transfer patients and the ones directly arriving to the emergency department (ED)

Informed consent forms (ICF) will be waived, as approved by the IRB.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with acute neurological symptoms suggestive of Stroke, ischemic or hemorrhagic ("Code Stroke"), regardless of presence or absence of ﬁnal Stroke diagnosis.
* Subjects aged 22 years or older.
* NCCT performed for Code Stroke screening.
* If the patient does not have a hemorrhage, a CTA (head and neck, performed for Code Stroke screening) should also be performed.
* NCCT and CTA have been processed by Methinks AI software.

Exclusion Criteria:

● Subject imaging does not meet Image Acquisition and DICOM Tag Requirements

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive Code Stroke patients, aged 22 or older, regardless of presence or absence of ultimate diagnosis of Ischemic Stroke or Hemorrhagic Stroke.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the sensitivity and specificity of the following Methinks AI modules: | Baseline, pre-intervention (Code Stroke presentation and screening), During Code Stroke treatment, Immediately After the stroke treatment, Up to Discharge or 7 Days (whichever is sooner).
  1. Methinks NCCT algorithm detecting ICA, M1, and M2 occlusions.
  2. Methinks NCCT algorithm detecting ICHs.
  3. Methinks CTA algorithm detecting ICA, M1, and M2 occlusions.

SECONDARY OUTCOMES:
Time Potential time reduction - difference in speed to LVO notification between Methinks NCCT-LVO and competitor CTA-LVO. | Baseline, pre-intervention (Code Stroke presentation and screening), During Code Stroke treatment, Immediately After the stroke treatment, Up to Discharge or 7 Days (whichever is sooner).
Time for NCCT-LVO Notification. | Baseline, pre-intervention (Code Stroke presentation and screening), During Code Stroke treatment, Immediately After the stroke treatment, Up to Discharge or 7 Days (whichever is sooner).
User experience. | 1 day (Questionnaire completed at individual site enrollment completion.)
  Site Principal Investigator will complete questionnaire based upon experience with use of the Methinks software and application.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — https://www.methinks.ai/